CLINICAL TRIAL: NCT02497560
Title: A Randomized Double Blind Placebo-Controlled Study To Investigate The Effect Of A Natural Dietary Supplement On Peri-Menopausal Symptoms
Brief Title: A Study To Investigate The Effect Of A Natural Dietary Supplement On Peri-Menopausal Symptoms
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Role of calcium in menopause is not clear. Product maybe reformulated and the study relaunched.
Sponsor: Physician Recommended Nutriceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PRN 20144
Record Dates: First submitted 2015-07-06; First posted 2015-07-14 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Menopause

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- Treatment (Active Comparator): all natural dietary supplement
  Interventions: Dietary Supplement: proprietary formula
- Treatment + Omega-3s (Other): all natural dietary supplement + omega-3s
  Interventions: Dietary Supplement: proprietary formula
- Placebo (Placebo Comparator): vegetable oil
  Interventions: Dietary Supplement: proprietary formula

INTERVENTIONS:
Dietary Supplement: proprietary formula

SUMMARY:
This is a randomized, masked, placebo controlled study to assess the effect on a nutritional dietary supplement on menopausal signs and symptoms in perimenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Age group between 45 and 65 at the time of informed consent.
* Physician diagnosis of menopause.
* History of substantial hot flashes > 4 episodes /day for last 2 weeks.
* Being post-menopausal with an intact uterus.
* Subject has provided signed and dated written informed consent before admission to the study.

Exclusion Criteria:

* Concurrent hot flash therapies (prescription medications including hormone replacement therapies, gabapentin or over the counter supplements), vaginal hormonal products (rings, creams, gels) or transdermal estrogen or estrogen/progestin products for 30 days before screening visit.
* Women currently or previously on anticoagulants, Vitamin K antagonists like warfarin in the past 3 months, or expected to be on anticoagulants in the near future.
* Women involved in other clinical studies within the last 30 days.
* Any women who, in the opinion of the principal investigator, is at poor medical or psychiatric risk for the study.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-03; Primary Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Hot flashes episodes | 12 weeks
  Diary

SECONDARY OUTCOMES:
Work productivity | 12 weeks
  Questionnaire
Quality of Life | 12 weeks
  Questionnaire

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Comprehensive Women's Care, Colorado Springs, Colorado
  - Dittrich Clinic, Philadelphia, Pennsylvania